CLINICAL TRIAL: NCT01757418
Title: Phase 1-2 Trial of Gamunex (Intravenous Gammaglobulin) for Sickle Cell Acute Pain
Brief Title: Intravenous Gammaglobulin for Sickle Cell Pain Crises
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: Food and Drug Administration (FDA) (U.S. Federal Agency); Case Western Reserve University (Other); Grifols Therapeutics LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 09-06-172; FD-R-005341-01 (Other Grant/Funding Number: FDA, OOPD); NCT00644865 (obsolete NCT alias)
Record Dates: First submitted 2012-11-08; First posted 2012-12-31 (Estimated); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Sickle Cell Disease; Pain
Keywords: Sickle Cell Disease; Pain; Immune Globulin
MeSH Terms: conditions — Anemia, Sickle Cell; Pain | interventions — gamma-Globulins; Immunoglobulins, Intravenous; Saline Solution

STUDY DESIGN:
Intervention Model Description: 1:1 randomization
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Intravenous Immune Globulin (IVIG) (Experimental): IVIG used in the trial is the GAMUNEX brand, at doses up through 800 mg/kg in Phase 1 and at 400mg/kg in Phase 2.
  Interventions: Drug: Immune Globulin Intravenous (IVIG)
- Normal saline (Placebo Comparator): An equivalent volume (weight-based) of normal saline
  Interventions: Other: Normal saline

INTERVENTIONS:
Drug: Immune Globulin Intravenous (IVIG) — A single dose of intravenous immune globulin or saline placebo administered within 24 hours of hospital presentation. The maximum dose in Phase I was 800 mg/kg. The dose for Phase II is 400mg/kg.
  Other Names: GAMUNEX (Talecris Biotherapeutics)
  Arms: Intravenous Immune Globulin (IVIG)
Other: Normal saline — A single dose of normal saline administered within 24 hours of hospital admission for uncomplicated pain crisis.
  Other Names: Placebo
  Arms: Normal saline

SUMMARY:
The purpose of this study is to determine whether intravenous immune globulin is safe and effective in the acute treatment of pain crises in sickle cell disease.

Funding Source: Food and Drug Administration (FDA), Office of Orphan Products Development (OOPD)

DETAILED DESCRIPTION:
Patients will be randomized to a single dose of IVIG versus normal saline placebo during an uncomplicated pain crisis. Length of VOC and other secondary endpoints will be monitored.

Phase 1: To determine the tolerability and obtain preliminary data on the clinical efficacy of IVIG treatment in a randomized, double-blind, placebo-controlled, dose escalation phase I clinical study of sickle cell disease patients admitted for acute vaso-occlusive crisis.

Phase II: To evaluate the effect of a single dose of 400mg/kg of IV Gamunex on length of VOC in subjects 8-14 years of age hospitalized for sickle cell VOC in a randomized, double blind placebo-controlled Phase 2 trial. To further evaluate safety of a single dose of 400mg/kg of IV Gamunex in subjects 8-14 years of age hospitalized for sickle cell VOC

ELIGIBILITY:
Each subject must fulfill each of the following Inclusion/Exclusion criteria at screening and continue to fulfill these criteria prior to dosing:

Inclusion Criteria:

* Documented Sickle Cell Disease (SS or S-β thalassemia genotype)
* Age 12-65 years for Phase 1 (Completed), 6-13.99 years for Phase 2 (Ongoing)
* Normal stroke risk as assessed by transcranial Doppler (TCD). A normal TCD in subjects 16 years of age and younger within the year prior to study drug administration are required
* Uncomplicated acute vaso-occlusive crisis requiring hospital admission and parenteral narcotic analgesics
* If prescribed Voxelotor: Consistent daily use of voxelotor in the past week AND able to continue Voxelotor inpatient OR no reported use in prior week

Exclusion Criteria:

* Concomitant acute process, including acute chest syndrome, potential serious infection, or clinically significant bleeding
* Fever > 38.5° C and clinical suspicion of infection
* Serum alanine aminotransferase >4x Upper Limit of Normal (ULN)
* Serum creatinine ≥1.3 mg/dL (or > than 95th percentile for age) or >300 mg/dL protein in spot urinalysis
* Known condition associated with renal dysfunction including but not limited to diabetes mellitus, uncontrolled hypertension, multiple myeloma, and congestive heart failure
* Any clinical evidence of prior stroke
* Prior thromboses or current estrogen use
* Current estrogen use
* Hb < 5 g/dL or > 10 g/dL
* Known Immunoglobulin A (IgA) deficiency or known allergy to gamma globulin
* Pregnancy or breastfeeding
* Current participation in another investigational drug study
* Current enrollment in a hypertransfusion program
* Previous participation in current study less than 3 months ago
* Current treatment with chronic transfusion
* Vaccination with a live attenuated virus in the preceding 6 weeks
* Documented history of illicit (e.g., heroin, cocaine) drug abuse
* Subject is otherwise not an appropriate study candidate, in the investigator's judgement, such as concern for opioid addiction or comorbid psychiatric diagnoses that may contribute to secondary gain in prolonged use of opioids or hospital stay
* Greater than 24 hours from time of presentation to the hospital for VOC
* Atrial fibrillation
* Right to left cardiac shunting due to patent foramen ovale or other anatomic cause
* Known magnetic resonance imaging/angiography (MRI/A) evidence of stroke or clinically significant central nervous system (CNS) vasculopathy at any age (Imaging done if clinically indicated)

Ages: 6 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2008-11; Primary Completion 2024-12-18 (Actual); Study Completion 2024-12-18 (Actual)

PRIMARY OUTCOMES:
Length of vaso-occlusive crisis (VOC) | Number of days from time of presentation to emergency room to end of crisis, average 4 days and maximum 30 days
  Length (duration) of vaso-occlusive crisis as measured from the time of presentation to the emergency room to end of VOC defined as 12 hours from the last dose of parenteral opioid analgesia for the treatment of VOC prior to hospital discharge. Group results will be summarized in number of days using univariate statistics.

SECONDARY OUTCOMES:
Total Opioid Use | From study drug infusion to end of crisis, average 4 days and maximum 30 days
  The total intravenous morphine equivalent use from the end of infusion to discharge will be compared between the IVIG and placebo group. This will require conversion of total amount of different opioids to the equivalent amounts of IV morphine in milligrams. Standard tables for equianalgesic opioid dosing will be used for these conversions. These tables account for opioid type, route of administration, and incomplete cross-tolerance, as needed, and are adjusted for body weight. Group results will be summarized in milligrams of opioid per kilogram of body weight (mg/kg) using univariate statistics.
Time to end of vaso-occlusive crisis | Number of days from start of study drug infusion to end of crisis, average 4 days and maximum 30 days
  Time to end of vaso-occlusive crisis as measured from start of study drug infusion to end of VOC end of VOC defined as 12 hours from the last dose of parenteral opioid analgesia for the treatment of VOC prior to hospital discharge. Group results will be summarized in number of days using univariate statistics.
Length of Hospitalization | From admission to discharge, average 4 days and maximum 30 days
  Length (duration) of Hospitalization will be summarized by study arm in months/days using univariate statistics.
Change in Macrophage-1 Antigen (Mac-1) expression | From Pre-infusion to 24-hours post-infusion
  Change in Mac-1 expression levels from prior to infusion to 24 hours following infusion will be assessed by the appropriate in vitro adhesion assay to measure adhesion to cellular surfaces. Mac-1 is a cell surface receptor found on lymphocytes and leukocytes and serves as a marker for binding and adhesion. Mac-1 expression levels increase upon activation by inflammatory stimuli leading to a higher concentration of Mac-1 molecules on the cell's surface. Percentage change in Mac-1 from pre-infusion will be summarized by study arm using univariate statistics.
Change in Lactate Dehydrogenase (LDH) levels | From Pre-infusion to 24-hours post-infusion
  Change in LDH levels from prior to infusion to 24 hours following infusion will be assessed. Percentage change in LDH concentration (in U/L) from pre-infusion will be summarized by study arm using univariate statistics. While normal LDH ranges vary by age/gender and thresholds have not been established for this study, higher LDH levels may serve as inflammatory biomarkers of hemolysis in patients with sickle cell disease and also be indicators of acute or chronic tissue damage.
Change in Hemoglobin (Hb) levels | From Pre-infusion to 24-hours post-infusion
  Change in Hb levels from prior to infusion to 24 hours following infusion will be assessed. Percentage change in Hb concentration (in g/dL) from pre-infusion will be summarized by study arm using univariate statistics. While normal Hb ranges vary by age/gender and thresholds have not been established for this study, in patients with sickle cell disease, decreased Hb levels may be indicative of anemia, increased risk of thromboembolic events, and organ and tissue damage.
Change in High-sensitivity C-reactive protein (hsCRP) levels | From admission to 24-hours post-infusion, average 4 days
  Change in hsCRP levels from admission to 24 hours following infusion will be assessed. Percentage change in hsCRP concentration (in mg/L) from admission will be summarized by study arm using univariate statistics. hsCRP serves a biomarker for inflammation. While normal ranges for hsCRP vary by age/gender and thresholds have not been established for this study, higher hsCRP levels may serve as a laboratory correlate of hospitalizations for pain or vaso-occlusive events in patients with sickle cell disease.
Rate of transfer to Intensive Care Unit (ICU) | From admission to discharge, average 4 days and maximum 30 days
  The percentage of patients who are admitted to the hospital's ICU for an emergent condition will be summarized by study arm.
Diagnosis leading to transfer to the ICU | From admission to discharge, average 4 days and maximum 30 days
  Diagnoses leading to transfer to the ICU will be summarized by study arm.
Number and type of Transfusions | From study drug infusion to discharge, average 4 days and maximum 30 days
  The number and types of intervening packed red blood cell transfusions administered during the study will be summarized by study arm. Types of red blood cell transfusions will be categorized (e.g., acute, intermittent, chronic, simple, exchange) and will be administered as clinically indicated and ordered by the physician in accordance with NIH-NHLBI evidence-based management of sickle cell disease guidelines.

CONTACTS AND LOCATIONS:
Overall Officials: Kerry Morrone, MD, Principal Investigator — Albert Einstein College of Medicine
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chang J, Shi PA, Chiang EY, Frenette PS. Intravenous immunoglobulins reverse acute vaso-occlusive crises in sickle cell mice through rapid inhibition of neutrophil adhesion. Blood. 2008 Jan 15;111(2):915-23. doi: 10.1182/blood-2007-04-084061. Epub 2007 Oct 11. PMID 17932253
- [Background] Turhan A, Jenab P, Bruhns P, Ravetch JV, Coller BS, Frenette PS. Intravenous immune globulin prevents venular vaso-occlusion in sickle cell mice by inhibiting leukocyte adhesion and the interactions between sickle erythrocytes and adherent leukocytes. Blood. 2004 Mar 15;103(6):2397-400. doi: 10.1182/blood-2003-07-2209. Epub 2003 Nov 20. PMID 14630831
- [Background] Shi PA, Manwani D, Olowokure O, Nandi V. Serial assessment of laser Doppler flow during acute pain crises in sickle cell disease. Blood Cells Mol Dis. 2014 Dec;53(4):277-82. doi: 10.1016/j.bcmd.2014.04.001. Epub 2014 May 21. PMID 24857171
- [Background] Manwani D, Frenette PS. Vaso-occlusion in sickle cell disease: pathophysiology and novel targeted therapies. Blood. 2013 Dec 5;122(24):3892-8. doi: 10.1182/blood-2013-05-498311. Epub 2013 Sep 19. PMID 24052549
- [Background] Manwani D, Chen G, Carullo V, Serban S, Olowokure O, Jang J, Huggins M, Cohen HW, Billett H, Atweh GF, Frenette PS, Shi PA. Single-dose intravenous gammaglobulin can stabilize neutrophil Mac-1 activation in sickle cell pain crisis. Am J Hematol. 2015 May;90(5):381-5. doi: 10.1002/ajh.23956. Epub 2015 Apr 1. PMID 25616042
- [Background] Manwani D, Xu C, Lee SK, Amatuni G, Cohen HW, Carullo V, Morrone K, Davila J, Shi PA, Ireland K, Keenan J, Frenette PS. Randomized phase 2 trial of Intravenous Gamma Globulin (IVIG) for the treatment of acute vaso-occlusive crisis in patients with sickle cell disease: Lessons learned from the midpoint analysis. Complement Ther Med. 2020 Aug;52:102481. doi: 10.1016/j.ctim.2020.102481. Epub 2020 Jun 9. PMID 32951731
- [Background] Jang JE, Hidalgo A, Frenette PS. Intravenous immunoglobulins modulate neutrophil activation and vascular injury through FcgammaRIII and SHP-1. Circ Res. 2012 Apr 13;110(8):1057-66. doi: 10.1161/CIRCRESAHA.112.266411. Epub 2012 Mar 13. PMID 22415018